CLINICAL TRIAL: NCT00357487
Title: Sentinel Lymph Node Identification in Case of Breast Cancer. Clinical Evaluation of a New Intra-operative Probe and a Mini Gamma Camera
Brief Title: Evaluation of Two New Medical Instruments Dedicated to the Sentinel Lymph Node Technique in Case of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Louis Pasteur University, Strasbourg (Other); Institut Pluridisciplinaire Hubert Curien, Strasbourg (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3704
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: Sentinel lymph node; Breast cancer; Lymphoscintigraphy; Probe; Operative gamma camera; Breast cancer and sentinel lymph node biopsy; Use of lymphoscintigraphy; Use of intraoperative gamma camera; Use of intraoperative probe
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Device: peroperative scintillating probe
Device: operative gamma camera

SUMMARY:
This project consists on the realization followed by the clinical validation of two medical instruments dedicated to the precise sentinel lymph nodes identification and localization in the case of breast cancer: an intra operative probe and an operative mini gamma camera. The sentinel lymph node technique, based on the propagation of cancer cells in the lymphatic system, allows a better evaluation of tumor staging, prognosis and therapeutic strategy determination. The goal of these instruments designed by physicians and physicists is to significantly improve the detection efficiency of the technique in order to reduce the false negative rate and then the recurrence risk, as well as the operative morbidity.Clinical oncologist surgeons and fundamental physics applied to medical imaging researchers are involved in this project. The clinical validation of the medical instruments will be organized in the Gynaecologic and Obstetric department of the Hospices Civils de Strasbourg with a series of 25 patients in the framework of a regular french protocol of clinical research.

ELIGIBILITY:
Inclusion Criteria:

* infiltrative breast cancer
* no suspect axillary lymph node
* no previous radiotherapy
* no previous chemotherapy
* no previous breast surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2006-06; Study Completion 2007-12

PRIMARY OUTCOMES:
The day before the surgery: Lymphoscintigraphy in a Nuclear Medicine Department
The day of the surgery: Preoperative axillary area mapping with the operative gamma camera. Search of sentinel lymph nodes with the probe
Post operative axillary area imaging with the operative gamma camera.

SECONDARY OUTCOMES:
Depth of the sentinel lymph nodes by a ruler before their excisions.
Radioactivity of the sentinel lymph nodes after their excisions.

CONTACTS AND LOCATIONS:
Overall Officials: Carole Mathelin, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Gyynécologie-Obstétrique -Hôpital Civil, Strasbourg, France

REFERENCES:
- [Derived] Mathelin C, Salvador S, Bekaert V, Croce S, Andriamisandratsoa N, Liegeois P, Prados E, Guyonnet JL, Grucker D, Brasse D. A new intraoperative gamma camera for the sentinel lymph node procedure in breast cancer. Anticancer Res. 2008 Sep-Oct;28(5B):2859-64. PMID 19031925
- [Derived] Mathelin C, Salvador S, Croce S, Andriamisandratsoa N, Huss D, Guyonnet JL. Optimization of sentinel lymph node biopsy in breast cancer using an operative gamma camera. World J Surg Oncol. 2007 Nov 17;5:132. doi: 10.1186/1477-7819-5-132. PMID 18021418